CLINICAL TRIAL: NCT05019326
Title: A Two-stage Adaptive Randomized Controlled Trial of Andrographis Paniculata Extract, Boesenbergia Rotunda Extract, and Standard Treatment in Asymptomatic COVID-19 Patients
Brief Title: Andrographis Paniculata vs Boesenbergia Rotunda vs Control in Asymptomatic COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MURA2021/652
Record Dates: First submitted 2021-08-21; First posted 2021-08-24 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Treatment; Andrographis; Boesenbergia; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Andrographis paniculata extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Andrographis extract (Experimental): Andrographis extract, equivalent to andrographolide 20 mg per capsule, for a total of 180 mg of andrographolide per day, dosing into 3 capsules taking before meal for 3 times per day, for 5 days.
  Interventions: Drug: Andrographis Paniculata
- Boesenbergia extract (Experimental): Boesenbergia extract, equivalent to pinostrobin 30 mg per capsule, for a total of 180 mg of pinostrobin per day, dosing into 2 capsules taking after meal for 3 times per day for 5 days.
  Interventions: Drug: Boesenbergia
- Standard supportive treatment (Other): Standard supportive treatment, as recommended by guideline from Ministry of Public Health, Thailand, there will be no antivirus given in this asymptomatic group
  Interventions: Other: Standard supportive treatment

INTERVENTIONS:
Drug: Andrographis Paniculata — Andrographis extract, equivalent to andrographolide 20 mg per capsule, for a total of 180 mg of andrographolide per day, dosing into 3 capsules taking before meal for 3 times per day, for 5 days.
  Arms: Andrographis extract
Drug: Boesenbergia — Boesenbergia extract, equivalent to pinostrobin 30 mg per capsule, for a total of 180 mg of pinostrobin per day, dosing into 2 capsules taking after meal for 3 times per day for 5 days.
  Arms: Boesenbergia extract
Other: Standard supportive treatment — as recommended by guidelines from the Ministry of Public Health, Thailand. No antivirus was given.
  Arms: Standard supportive treatment

SUMMARY:
The purpose of this study is to examine the effect of Andrographis Extract, Boesenbergia Extract compared to standard treatment in asymptomatic COVID patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 60 years old
2. Have been diagnosed as new COVID-19 case by RT-PCR since disease onset to admission less than 7 days
3. Have asymptomatic infection assessed by the World Health Organization (WHO) disease category
4. Do not have any of following disease or conditions

   1. Body weight > 90 kg or BMI > 30 kg/m2
   2. Hypertension that needs antihypertensive medication
   3. Diabetes
   4. Cardiovascular diseases including congenital heart disease
   5. Cerebrovascular diseases
   6. Chronic kidney and chronic liver diseases
   7. COPD or chronic lung diseases
   8. Lymphocyte <1,000 cells/mm3
   9. Late-stage cancer
   10. Auto-immune disease (e.g., SLE, Rheumatoid arthritis, multiple sclerosis, etc.) or currently on immunosuppressive drug
   11. Coagulation disorders or platelet disorders and are being treated with anticoagulants such as warfarin, clopidogrel
   12. Pregnancy
5. Willing to participate with the study and sign inform consents.

(Withdrawal criteria)

1. Patients withdraw from the study
2. Have severe adverse effect that may relate to Andographolide or Boesenbergia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3060 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Require hospitalization in the hospital | 28 days
  From WHO clinical progression scale (0-10):
  0: Uninfected with no viral RNA detected
  1. Asymptomatic with viral RNA detected
  2. Symptomatic and independent
  3. Symptomatic with assistance needed
  4. Hospitalized with no oxygen therapy needed
  5. Hospitalized with oxygen mask or nasal prongs
  6. Hospitalized with oxygen by NIV or high flow
  7. Intubation and mechanical ventilation with pO2/FiO2 >= 150 or SpO2/FiO2 >= 200
  8. Mechanical ventilation with pO2/FiO2 < 150 (SpO2/FiO2 <200) or vasopressor
  9. Mechanical ventilation with pO2/FiO2 < 150 and vasopressor, dialysis, or ECMO
  10. Dead
  Outcome 4 or more considered as hospitalization

SECONDARY OUTCOMES:
Individual status from WHO clinical progression scale (0-10) | 28 days
  From WHO clinical progression scale:
  0: Uninfected with no viral RNA detected
  1. Asymptomatic with viral RNA detected
  2. Symptomatic and independent
  3. Symptomatic with assistance needed
  4. Hospitalized with no oxygen therapy needed
  5. Hospitalized with oxygen mask or nasal prongs
  6. Hospitalized with oxygen by NIV or high flow
  7. Intubation and mechanical ventilation with pO2/FiO2 >= 150 or SpO2/FiO2 >= 200
  8. Mechanical ventilation with pO2/FiO2 < 150 (SpO2/FiO2 <200) or vasopressor
  9. Mechanical ventilation with pO2/FiO2 < 150 and vasopressor, dialysis, or ECMO
  10. Dead
  More on the scale - worse outcome
Pneumonia | 28 days
  Pneumonia by diagnosis or chest radiography
Quality of life by EQ5D-5L | 28 days
  Quality of life by EQ5D-5L
  Scale of 0 to 100 for overall health state (lower is worse) and 1 to 5 in each of 5 domains. (higher score is worse)
Side effect of medication | 28 days
  Renal and liver function elevation and other anticipated/unanticipated side effect:
  Side effect of medication will be classified according to common terminology criteria for adverse events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
May shared IPD upon sponsor decision.